CLINICAL TRIAL: NCT06966219
Title: Impact of Trigger Protocol on the Rate of Pregnancy After Intracytoplasmic Sperm Injection: A Prospective Cohort Study
Brief Title: Trigger Protocol on the Rate of Pregnancy After Intracytoplasmic Sperm Injection
Status: Active, not recruiting | Type: Observational
Sponsor: Suez University (Other)
Responsible Party: Principal Investigator, Ahmed Sewidan, lecturer of obstetrics and gynecology, Suez University
Other Study IDs: 3
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Infertility
Keywords: icsi; dual trigger
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Ninety women presenting with infertility were recruited from the outpatient clinic. Baseline data, including demographic and medical history, BMI, and laboratory investigations (CBC, renal and liver function tests, coagulation profile along with hormonal profile ), were collected. All patients underwent intracytoplasmic sperm injection for infertility.
  Interventions: Other: Intracytoplasmic sperm injection

INTERVENTIONS:
Other: Intracytoplasmic sperm injection — • All patients will commence controlled ovarian hyperstimulation (COH) on day 2 or 3 of their menstrual cycle. The initial treatment will be a daily administration of either highly purified human menopausal gonadotropin (hMG) or recombinant FSH (rFSH, Gonal-F 150 IU, Merck Serono, S.P.A, Italy) administered subcutaneously and intramuscularly for a duration of 10-12 days. The treatment will be continued until the final oocyte maturation. The starting dosage will be tailored based on the patient's age, antral follicle count (AFC), body mass index (BMI), serum FSH and AMH levels on days 2-3, as well as the patient's previous response to COH.

SUMMARY:
Infertility is a condition affecting both female and male, characterized by the inability to conceive after 12 months or more of regular, unprotected sexual activity. All over the world, over 186 million people are affected by this condition, with the majority living in developing countries. In developing countries, the prevalence of infertility among women of reproductive age is estimated to affect one in every four couples. Type of the trigger during intracytoplasmic sperm injection might has impact on pregnancy rate.

DETAILED DESCRIPTION:
When 3rd generation Gonadotropin-releasing hormone antagonists (GnRH-a) were introduced in the 1990s for ovarian induction protocols, it became possible to trigger final oocyte maturation and ovulation with a single bolus of GnRH-a as an alternative to Human chorionic gonadotropin (HCG). Although some studies have suggested an increase in the percentage of mature 2 ((MII) oocytes retrieved with GnRH-a compared to HCG, it has been found that triggering ovulation with only GnRH agonist leads to a suboptimal luteal phase. The term "dual trigger" was first defined as the combination of a GnRH agonist and a low dose of HCG for triggering terminal oocyte maturation and avoid ovarian hyperstimulation syndrome (OHSS) in GnRH antagonist protocols.

Lin et al, conducted a retrospective study represent normal responders undergoing intracytoplasmic sperm injection )ICSI (with a GnRH antagonist trigger. They demonstratedsignificant improvements in the total number of retrieved oocytes, the number of mature (MII) oocytes, and rates of embryo implantation, clinical pregnancy, ongoing pregnancy, and live birth rate when the dual trigger protocol was used. Similarly, Lu et al. presented a retrospective analysis of fertility centers records where final oocyte maturation was triggered by either GnRH alone (Decapeptyl 0.1-0.2 mg) or in combination with HCG (1,000, 2,000, or 5,000 IU). They concluded that employing a dual trigger with a low dose of hCG (1,000 IU) as an adjunct to GnRH-a significantly improved the oocyte retrieval rate in suboptimal responders.

ELIGIBILITY:
Inclusion Criteria:

• Patients are less than 38 years old

* Patients have primary or secondary infertility
* Patient is candidate for ICSI
* Normal antral follicles count
* AMH more than 1

Exclusion Criteria:

* Age more than 38 years old
* Patients have other options for assisted reproductive techniques like
* intrauterine insemination.
* Severe male factor
* AMH less than 1
* Recurrent ICSI failure

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: females attended the clinic with a history of infertility required Intracytoplasmic sperm inaction
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate after dual versus single trigger during ICSI | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wessam aboelghar, Principal Investigator — faculty of medicine, Suez university Suez, Suez, Egypt
Locations (1):
- faculty of medicine, Suez university, Suez, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin MH, Wu FS, Lee RK, Li SH, Lin SY, Hwu YM. Dual trigger with combination of gonadotropin-releasing hormone agonist and human chorionic gonadotropin significantly improves the live-birth rate for normal responders in GnRH-antagonist cycles. Fertil Steril. 2013 Nov;100(5):1296-302. doi: 10.1016/j.fertnstert.2013.07.1976. Epub 2013 Aug 28. PMID 23993928
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Thomas S. Gonadotropin-releasing hormone agonist combined with a reduced dose of human chorionic gonadotropin for final oocyte maturation in fresh autologous cycles of in vitro fertilization. Fertil Steril. 2008 Jul;90(1):231-3. doi: 10.1016/j.fertnstert.2007.06.030. Epub 2007 Nov 5. PMID 17981269
- [Background] Segal S, Casper RF. Gonadotropin-releasing hormone agonist versus human chorionic gonadotropin for triggering follicular maturation in in vitro fertilization. Fertil Steril. 1992 Jun;57(6):1254-8. PMID 1601147
- [Background] Humaidan P, Westergaard LG, Mikkelsen AL, Fukuda M, Yding Andersen C. Levels of the epidermal growth factor-like peptide amphiregulin in follicular fluid reflect the mode of triggering ovulation: a comparison between gonadotrophin-releasing hormone agonist and urinary human chorionic gonadotrophin. Fertil Steril. 2011 May;95(6):2034-8. doi: 10.1016/j.fertnstert.2011.02.013. Epub 2011 Mar 5. PMID 21377153
- [Background] Mascarenhas MN, Flaxman SR, Boerma T, Vanderpoel S, Stevens GA. National, regional, and global trends in infertility prevalence since 1990: a systematic analysis of 277 health surveys. PLoS Med. 2012;9(12):e1001356. doi: 10.1371/journal.pmed.1001356. Epub 2012 Dec 18. PMID 23271957